CLINICAL TRIAL: NCT00733798
Title: A Phase 1/2, Multi-Center, Safety and Efficacy Study Evaluating Intravenously Administered 131I-TM601 in Patients With Progressive and/or Recurrent Malignant Melanoma
Brief Title: A Safety and Efficacy Study of Intravenous 131I-TM601 in Adult Patients With Malignant Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: For Strategic Reasons
Sponsor: TransMolecular (Industry)
Responsible Party: Susan Stewart, TransMolecular
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TM601-011
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2009-05-11 (Estimated); Status verified 2009-05

CONDITIONS: Melanoma; Malignant Melanoma; Metastatic Melanoma
Keywords: Melanoma; Malignant melanoma; metastatic melanoma; Phase 1; Phase 2
MeSH Terms: conditions — Melanoma | interventions — Chlorotoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: 131I-TM601

INTERVENTIONS:
Drug: 131I-TM601 — After a single 20mCi/0.4 mg Imaging Dose of 131I-TM601, patients in the Dose Escalation Phase will be administered between 2-5 weekly doses of 131I-TM601 at 1.2 mCi/kg of lean body mass (specific activity of 131I-TM601 will be maintained at 50 mCi 131I/mg TM601 for all doses administered in this study.) Patients in the Efficacy Phase of the study will be treated at the Maximum Tolerated Dose established in the Dose Escalation Phase.
  Other Names: chlorotoxin

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of 131I-TM601 in the treatment of adult patients with progressive and/or recurrent malignant melanoma.

DETAILED DESCRIPTION:
This is a multi-center, Phase 1/2 study evaluating the use of multiple intravenous doses of 131I-TM601 in adults patients with progressive and/or recurrent malignant melanoma (Stage IIIc or IV) with measurable disease who have failed first line/standard therapy.

The study will be conducted in 2 phases. During the first, Dose Escalation Phase, eligible patients wil be assigned in groups of 3-6 (depending upon the treatment response seen at each dose) to dose cohorts of between 2-5 weekly IV doses of 131I-TM601. Escalation to the next highest dose during the Dose Escalation Phase will be dependent upon demonstrated tolerance in the previous dosing group. In the second, Efficacy Phase, all patients will be treated with the Maximum Tolerated Dose determined in the Dose Escalation Phase.

Prior to initiating treatment, all patients will be administered a single imaging dose of 131I-TM601, IV, as an Imaging Dose to evaluate tumor uptake. Only patients demonstrating tumor uptake will remain on the study.

Patients in both study phases will have safety parameters evaluated continuously throughout the study. Clinical response to 131I-TM601 will be assessed in each study patient at 28 days following the final study dose, and then at 2-month intervals, starting at 3 months following the first study dose (during the first year of follow-up), and finally at 3-month intervals thereafter until disease progression.

ELIGIBILITY:
Inclusion Criteria:

Patient MUST:

1. Have signed and dated written informed consent.
2. Be aged ≥ 18 years old at time of informed consent.
3. Have histologically proven Stage IIIc or IV malignant melanoma with documented progression during or following the most recent prior melanoma therapy.
4. Have measurable disease, defined as lesions that can be accurately measured in at least one dimension as > 20 mm with conventional techniques (CT) or > 10 mm with spiral CT scan or brain MRI.
5. Have failed at least 1 prior therapy for melanoma or refused first-line, standard therapy.
6. Have an ECOG performance status of 0 - 1.
7. Have a life expectancy, based on the Investigator's judgment, of > 3 months.
8. On screening ECG, have a QTc interval of < 450 ms.
9. If taking steroids, be on a dose that is stable for at least 5 days prior to the Imaging Dose.
10. Have recovered from the toxicity of all previous therapy prior to enrollment. If the patient has undergone recent major surgery, an interval of at least 3 weeks must have elapsed between the surgery and the date of the Imaging Dose.
11. Have acceptable laboratory results as follows:

    1. Hemoglobin ≥ 9g/dL
    2. ANC ≥ 1,500 mm3
    3. Platelet count ≥ 150,000 mm3
    4. PT <1.5 ULN
    5. PTT < 1.5 ULN
    6. Total Bilirubin < 2.0 mg/dL
    7. AST/ALT < or = 5 ULN
    8. Serum Creatinine < or = 2 mg/dL
12. Have a negative serum pregnancy test within 14 days of study drug administration, if female and of child bearing potential.
13. Agree to use an effective form of contraception to avoid pregnancy, if fertile (applicable to both male and female patients).
14. Agree to refrain from nursing, if female.
15. Be able to comply with treatment plan, study procedures, and follow-up examinations.

    If enrolled in the single site Sub-Study, patient MUST:
16. Have at least one accessible biopsy site and a second measurable target site per RECIST criteria.
17. Agree to pre-infusion and post-infusion biopsies of tumor lesions.

Exclusion Criteria:

Patient May Not:

1. Have a serious concurrent infection or medical illness which would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety. Examples of medical illnesses include, but are not limited to, the following: uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, known history of HIV, Hepatitis B or Hepatitis C infection, or psychiatric illness/social situation which would limit compliance with study requirements.
2. Have CNS metastases, unless, in the PI's judgment, the CNS involvement is stable and not likely to require further palliative therapy to the CNS during the course of the treatment protocol. If previous treatment has included radiotherapy, CNS disease should be stable at least 6 weeks from receipt of previous radiotherapy.
3. Have a prior malignancy with less than 3-year disease-free interval, except for adequately treated basal cell or squamous cell carcinoma of the skin, or in situ cancer of the cervix.
4. Have received radiation treatments < 6 weeks prior to first study drug administration (Imaging Dose).
5. Have previously received radiation to ≥ 25% red bone marrow.
6. Have received any cytotoxic chemotherapy, hormonal therapy, or immunotherapy, whether conventional or investigational, < 4 weeks prior to receiving the first study drug (Imaging Dose) administration in this study (6 weeks for mitomycin-C or nitrosoureas).
7. Have a history of pulmonary embolism within 1 year or deep venous thrombosis within six months of study enrollment.
8. Current or recent history of high-dose aspirin, warfarin, or heparin use (Aspirin < or = 81 mg/day, low-dose warfarin < 1 mg/day, or low-dose heparin for IV catheter patency is allowed).
9. Received investigational agents within 4 weeks prior to receiving the first study drug (Imaging Dose) administration in this study.
10. Have a history of allergic reactions attributed to compounds of similar chemical or biological composition to 131I-TM601 e.g. iodine or iodine-containing drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)

PRIMARY OUTCOMES:
Safety profile, as evaluated by incidence, severity, duration, causality, and seriousness of adverse events as well as by changes in patient's physical examination, vital signs, and clinical laboratory assessments. | duration of the study
6 month progression-free survival | duration of study

SECONDARY OUTCOMES:
Clinical response, time to disease progression, and overall survival. | duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gribbin, MD, Principal Investigator — Lacks Cancer Center; Neil Senzer, MD, Principal Investigator — Mary Crowley Cancer Center; Anna Pavlick, DO, Principal Investigator — New York University Cancer Center
Locations (3):
- United States (3):
  - Lacks Cancer Center, Grand Rapids, Michigan
  - New York University School of Medicine, New York, New York
  - Mary Crowley Cancer Center, Dallas, Texas

REFERENCES:
- [Background] Mamelak AN, Rosenfeld S, Bucholz R, Raubitschek A, Nabors LB, Fiveash JB, Shen S, Khazaeli MB, Colcher D, Liu A, Osman M, Guthrie B, Schade-Bijur S, Hablitz DM, Alvarez VL, Gonda MA. Phase I single-dose study of intracavitary-administered iodine-131-TM-601 in adults with recurrent high-grade glioma. J Clin Oncol. 2006 Aug 1;24(22):3644-50. doi: 10.1200/JCO.2005.05.4569. PMID 16877732
- [Background] Hockaday DC, Shen S, Fiveash J, Raubitschek A, Colcher D, Liu A, Alvarez V, Mamelak AN. Imaging glioma extent with 131I-TM-601. J Nucl Med. 2005 Apr;46(4):580-6. PMID 15809479
- [Background] Lyons SA, O'Neal J, Sontheimer H. Chlorotoxin, a scorpion-derived peptide, specifically binds to gliomas and tumors of neuroectodermal origin. Glia. 2002 Aug;39(2):162-73. doi: 10.1002/glia.10083. PMID 12112367
- [Background] Mamelak AN, Jacoby DB. Targeted delivery of antitumoral therapy to glioma and other malignancies with synthetic chlorotoxin (TM-601). Expert Opin Drug Deliv. 2007 Mar;4(2):175-86. doi: 10.1517/17425247.4.2.175. PMID 17335414